CLINICAL TRIAL: NCT06797999
Title: A First-in-human, Phase 1/2, Multicenter, Open-label, Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of ADCE-D01, a Humanized Anti-human uPARAP Antibody Linked to a Topoisomerase I Inhibitor, in Patients With Metastatic and/or Unresectable Soft Tissue Sarcoma
Brief Title: First-in-Human Study of ADCE-D01 in Soft Tissue Sarcoma
Acronym: ADCElerate1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adcendo ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCE-D01-001; 2024-516900-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Soft Tissue Sarcoma; Unresectable Soft Tissue Sarcoma
Keywords: Phase 1/Phase 2; Sequential; Treatment
MeSH Terms: conditions — Sarcoma | interventions — Immunoconjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCE-D01 (Other): ADCE-D01
  Interventions: Biological: Antibody-drug conjugate (ADC)

INTERVENTIONS:
Biological: Antibody-drug conjugate (ADC) — ADCE-D01 is an antibody-drug conjugate (ADC) composed of an anti-urokinase plasminogen activator receptor-associated protein (uPARAP) antibody, AB-004, conjugated to a topoisomerase I inhibitor, P1021, via a protease cleavage tetra-peptide linker.
  Other Names: ADCE-D01

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and efficacy of ADCE-D01.

DETAILED DESCRIPTION:
Safety and Tolerability evaluated by incidence of DLTs. Efficacy evaluated by antitumor activity; ORR, DOR, PFS, CBR and TTR per RECIST v i.1.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Histologically confirmed STS with metastatic and/or unresectable disease (not amenable to treatment with curative intent).
3. Prior treatment with at least one but no more than two lines of cytotoxic systemic therapy for metastatic/unresectable disease.
4. Measurable disease as per RECIST v 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of at least 3 months.
7. A male patient must agree to use barrier contraception during the treatment period and for at least 4 months after the last infusion of study treatment, and refrain from donating sperm during this period. Male patients with a pregnant partner must practice sexual abstinence or use a barrier method of contraception (e.g., condom) to prevent exposure of the fetus or neonate.
8. A female patient is eligible if not pregnant, not breast feeding, and not a woman of childbearing potential (WOCBP), or agrees to follow the contraceptive guidance during the treatment period and for at least 7 months after last infusion of study treatment.

Exclusion Criteria:

1. Patients who have had systemic anticancer therapy, including any investigational agent within 4 weeks or 5 half-lives (whichever is shorter) prior to study treatment administration.
2. Primary brain malignancy or known, untreated central nervous system (CNS) or leptomeningeal metastases, or symptoms suggesting CNS involvement.
3. Clinically significant cardiovascular disease
4. Patients with acute infection with human immunodeficiency virus (HIV) 1 or HIV 2.
5. Current active liver disease due to hepatitis B
6. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on a chest computed tomography (CT) scan at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2029-02-27 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD/maximum administered dose and RP2DS of ADCE-D01. | From enrollment to the end of Phase 1b (Approximately 18 months after enrollment)
  Measuring incidence of dose-limiting toxicities (DLTs)
Assess the safety and tolerability of ADCE-D01 | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Nature, incidence, severity and causality of treatment-emergent adverse events (TEAEs) and changes from baseline in laboratory parameters using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0).
  Tolerability as assessed by TEAEs leading to dose interruption, reduction and/or discontinuation.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Time to maximum plasma concentration will be assessed to inform ADCE-D01 PK profile
ADCE-D01 time to Cmax (Tmax) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Time to Cmax (Tmax) will be assessed to characterize the ADCE-D01 PK profile
ADCE-D01 area under the concentration-time curve (AUC) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  ADCE-D01 area under the concentration-time curve (AUC) will be assessed to characterize PK profile
Evaluate ADCE-D01 objective response rate (ORR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Objective response rate (ORR) per RECIST v1.1 by Investigator assessment
Evaluate ADCE-D01 duration of response (DOR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Duration of response DOR, measured per RECIST v1.1 by Investigator assessment will be used to further characterize the durability of tumor response of ADCE-D01
ADCE-D01 progression-free survival (PFS) | Throughout the trial duration, completion expected approximately 18 months from completed enrollmen
  Progression-free survival (PFS) assessed by Investigator per RECIST v1.1 to evaluate preliminary antitumor activity.
ADCE-D01 clinical benefit rate (CBR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  clinical benefit rate (CBR) assessed by Investigator per RECIST version 1.1 to evaluate preliminary antitumor activity of ADCE-D01
ADCE-D01 time to response (TTR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  time to response (TTR) assessed by Investigator per RECIST version 1.1 to evaluate preliminary antitumor activity of ADCE-D01

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Of Texas MD Anderson Cancer Center, Houston, Texas
- Universitair Ziekenhuis Leuven (UZ Leuven) - Campus Gasthuisberg, Leuven, Belgium
- Centre Léon Bérard, Lyon, France
- Universitätsklinikum Essen West German Tumor Center, Essen, Germany
- Royal Marsden, London, United Kingdom